CLINICAL TRIAL: NCT02812797
Title: Prognostic Value of Adipokine Levels of Patients With Chronic Heart Failure
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Dr, Chongqing Medical University
Other Study IDs: 2016-38-2
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Chronic Heart Failure
Keywords: Adipokines; Chronic Heart Failure; Prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether expressions of adipokines can provide prognostic information concerning patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are giving open chest surgical treatment with a history of chronic heart failure (NYHA II ~ IV) more than 6 months.
* Patients from whom informed consent has been properly obtained in writing prior to start of the trial.

Exclusion Criteria:

* Patients with concurrent infection or any documented inflammatory illness, such as arthritis or connective tissue diseases,or any other malignancy.
* Patients with a history of cardiomyopathy.
* Patients with Chronic arrhythmia.
* Pregnant women
* Severe hepatic dysfunction or End-stage renal failure.
* Uncontrolled hypertension.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Chronic Heart Failure
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Change from Baseline at 3, 6 and 12 months

SECONDARY OUTCOMES:
New York Heart Association (NYHA) Classification | Week:4
re-hospitalization | Change from Baseline at 3, 6 and 12 months
  Heart failure with re-hospitalization is documented by at least one of the following: worse exercise tolerance and respiratory distress with NYHA class III or IV symptoms, presence of pulmonary rales, or chest radiography showing pulmonary congestion, which needs an augmented decongestive regimen with oral or intravenous medications during an in-hospital stay.
plasma brain natriuretic peptide (BNP) concentration | Week:4
Cardiovascular death | Change from Baseline at 3, 6 and 12 months
Cardiac transplantation | Change from Baseline at 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, doctor, Study Director — Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided